CLINICAL TRIAL: NCT00878384
Title: A Randomised Trial to Assess Catheter Ablation Versus Rate-Control in the Management of Persistent Atrial Fibrillation in Chronic Heart Failure
Brief Title: Catheter Ablation Versus Medical Rate Control for Atrial Fibrillation in Patients With Heart Failure
Acronym: ARC-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008CI008B
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Atrial Fibrillation; Heart Failure
Keywords: Atrial Fibrillation; Heart Failure; Heart Rate Control; Catheter Ablation
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rate control (Active Comparator): Strategy of 'rate-control': acceptance of atrial fibrillation, and dose-adjusted drug therapy as needed to control ventricular rate.
  Interventions: Drug: Medication to control ventricular rate in AF
- Catheter Ablation (Active Comparator): Strategy of 'rhythm control' by catheter ablation: patients will undergo catheter ablation with the intention of restoring sinus rhythm.
  Interventions: Procedure: Catheter Ablation for Persistent Atrial Fibrillation

INTERVENTIONS:
Drug: Medication to control ventricular rate in AF — Standard pharmacologic rate control. Current therapy will be adjusted to achieve rate-control targets of <80bpm and <110bpm on exercise (6 minute walk). Where necessary, additional medication will be given as per standard practice (digoxin or beta-blocker). Typical does: Digoxin 62.5-250mcg o.d. ; Bisoprolol 1.25-20mg o.d.; Carvedilol 3.125-50mg b.d. ; Nebivolol 1.25-10mg o.d.
  Arms: Rate control
Procedure: Catheter Ablation for Persistent Atrial Fibrillation — Radiofrequency catheter ablation, which may include pulmonary vein isolation, atrial substrate modification, and/or linear ablation.
  Other Names: Radiofrequency catheter ablation; AF ablation; LA maze
  Arms: Catheter Ablation

SUMMARY:
It is still uncertain what the best treatment is for patients who have both atrial fibrillation (AF) and heart failure. The aim of the study is to help identify the optimal treatment for patients with these two significant medical conditions. This will be performed by comparing two alternative strategies for AF management: catheter ablation (to restore normal rhythm) and medical therapy (to control heart rate, but not aiming ro restore normal rhythm). After random assignment, the effect of each strategy will be assessed by looking for changes in exercise capacity, symptoms, heart pump function, and quality of life during 12 months of follow-up.

DETAILED DESCRIPTION:
Currently available evidence suggests that occurrence of AF in patients with heart failure (HF) leads to a decline in exercise tolerance, worsened quality of life, increased hospitalisation, and in many studies an increase in mortality. These may be explained by the haemodynamic effects of AF i.e. reduction in functional cardiac output due to inappropriate heart rates, irregularity, and loss of atrial contraction, plus the risk of thromboembolism.

Evidence from large clinical studies has shown that patients with heart failure fare better if sinus rhythm can be restored, but on the contrary a 'rhythm control' strategy (as intention to treat) of cardioversion or antiarrhythmic drugs to achieve sinus rhythm has not been shown to be superior to the strategy of rate control. These apparently contradictory findings might be explained by the poor efficacy and side effects associated with current rhythm control strategies, or could reflect that AF is merely a passive marker of underlying disease severity. However, many studies would point to the former, and it might be hypothesised that the theoretical benefits of sinus rhythm could be seen for real in clinical practice if a superior rhythm-control strategy was used.

Catheter ablation, a relatively new treatment for atrial fibrillation, has been shown to be feasible in a non-randomised heart failure patient cohort, with markers suggesting improvement of cardiac function.

This prospective clinical trial will enrol HF patients on optimal therapy, with documented persistent AF, and compare the strategies of catheter-ablation and medical rate control in a 1:1 randomised fashion.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years, < 80years
* NYHA II-IV symptoms
* Impairment of left ventricular systolic function (left ventricular ejection fraction estimated as ≤ 35% by radionuclide ventriculography)
* Documented AF lasting for at least 7 days (persistent or permanent AF)

Exclusion criteria:

* CRT or ICD device implanted in the previous 6 months
* AV nodal ablation within previous 3 months
* Prior AV nodal ablation or complete heart block with a single chamber pacemaker
* Contraindication to anticoagulation
* Persistent thrombus in the left atrium despite anticoagulation
* Active malignancy
* Cerebrovascular accident within the previous 6 months
* Reversible causes of AF including thyroid disorders, alcohol, recent surgery
* Reversible causes of heart failure including acute myocarditis or alcohol
* Cardiac events including myocardial infarction (MI), percutaneous coronary intervention (PCI), valve or coronary bypass surgery within the previous 3 months
* Prior AF ablation procedure
* Previous heart transplant, or on urgent heart transplant waiting list
* Severe neuro-muscular disease
* Creatinine clearance <30 ml/min
* Serum bilirubin >50 micromol/L
* Active participation in another research study
* Unable to understand and comply with protocol or give written informed consent
* Body mass index >35 (kg/m2)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-04; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Peak oxygen consumption at cardiopulmonary exercise test | 12 months

SECONDARY OUTCOMES:
Left ventricular ejection fraction | 12 months
Quality of Life score | 3, 6 and 12 months
6 minute walk distance | 3, 6 and 12 months
Level of plasma neurohormones (including BNP) | 3, 6 and 12 months
Freedom from AF | 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tom Wong, MD FESC, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton & Harefield NHS Trust, London, United Kingdom

REFERENCES:
- [Background] Hsu LF, Jais P, Sanders P, Garrigue S, Hocini M, Sacher F, Takahashi Y, Rotter M, Pasquie JL, Scavee C, Bordachar P, Clementy J, Haissaguerre M. Catheter ablation for atrial fibrillation in congestive heart failure. N Engl J Med. 2004 Dec 2;351(23):2373-83. doi: 10.1056/NEJMoa041018. PMID 15575053
- [Background] Dries DL, Exner DV, Gersh BJ, Domanski MJ, Waclawiw MA, Stevenson LW. Atrial fibrillation is associated with an increased risk for mortality and heart failure progression in patients with asymptomatic and symptomatic left ventricular systolic dysfunction: a retrospective analysis of the SOLVD trials. Studies of Left Ventricular Dysfunction. J Am Coll Cardiol. 1998 Sep;32(3):695-703. doi: 10.1016/s0735-1097(98)00297-6. PMID 9741514
- [Background] Middlekauff HR, Stevenson WG, Stevenson LW. Prognostic significance of atrial fibrillation in advanced heart failure. A study of 390 patients. Circulation. 1991 Jul;84(1):40-8. doi: 10.1161/01.cir.84.1.40. PMID 2060110
- [Background] Swedberg K, Olsson LG, Charlesworth A, Cleland J, Hanrath P, Komajda M, Metra M, Torp-Pedersen C, Poole-Wilson P. Prognostic relevance of atrial fibrillation in patients with chronic heart failure on long-term treatment with beta-blockers: results from COMET. Eur Heart J. 2005 Jul;26(13):1303-8. doi: 10.1093/eurheartj/ehi166. Epub 2005 Mar 14. PMID 15767288
- [Background] Roy D, Talajic M, Nattel S, Wyse DG, Dorian P, Lee KL, Bourassa MG, Arnold JM, Buxton AE, Camm AJ, Connolly SJ, Dubuc M, Ducharme A, Guerra PG, Hohnloser SH, Lambert J, Le Heuzey JY, O'Hara G, Pedersen OD, Rouleau JL, Singh BN, Stevenson LW, Stevenson WG, Thibault B, Waldo AL; Atrial Fibrillation and Congestive Heart Failure Investigators. Rhythm control versus rate control for atrial fibrillation and heart failure. N Engl J Med. 2008 Jun 19;358(25):2667-77. doi: 10.1056/NEJMoa0708789. PMID 18565859
- [Background] Pedersen OD, Brendorp B, Elming H, Pehrson S, Kober L, Torp-Pedersen C. Does conversion and prevention of atrial fibrillation enhance survival in patients with left ventricular dysfunction? Evidence from the Danish Investigations of Arrhythmia and Mortality ON Dofetilide/(DIAMOND) study. Card Electrophysiol Rev. 2003 Sep;7(3):220-4. doi: 10.1023/B:CEPR.0000012386.82055.81. PMID 14739717
- [Background] Corley SD, Epstein AE, DiMarco JP, Domanski MJ, Geller N, Greene HL, Josephson RA, Kellen JC, Klein RC, Krahn AD, Mickel M, Mitchell LB, Nelson JD, Rosenberg Y, Schron E, Shemanski L, Waldo AL, Wyse DG; AFFIRM Investigators. Relationships between sinus rhythm, treatment, and survival in the Atrial Fibrillation Follow-Up Investigation of Rhythm Management (AFFIRM) Study. Circulation. 2004 Mar 30;109(12):1509-13. doi: 10.1161/01.CIR.0000121736.16643.11. Epub 2004 Mar 8. PMID 15007003
- [Background] Hagens VE, Crijns HJ, Van Veldhuisen DJ, Van Den Berg MP, Rienstra M, Ranchor AV, Bosker HA, Kamp O, Tijssen JG, Veeger NJ, Van Gelder IC; RAte Control versus Electrical cardioversion for persistent atrial fibrillation study group. Rate control versus rhythm control for patients with persistent atrial fibrillation with mild to moderate heart failure: results from the RAte Control versus Electrical cardioversion (RACE) study. Am Heart J. 2005 Jun;149(6):1106-11. doi: 10.1016/j.ahj.2004.11.030. PMID 15976795
- [Derived] Jones DG, Haldar SK, Jarman JW, Johar S, Hussain W, Markides V, Wong T. Impact of stepwise ablation on the biatrial substrate in patients with persistent atrial fibrillation and heart failure. Circ Arrhythm Electrophysiol. 2013 Aug;6(4):761-8. doi: 10.1161/CIRCEP.113.000390. Epub 2013 Jul 23. PMID 23881779
- [Derived] Jones DG, Haldar SK, Hussain W, Sharma R, Francis DP, Rahman-Haley SL, McDonagh TA, Underwood SR, Markides V, Wong T. A randomized trial to assess catheter ablation versus rate control in the management of persistent atrial fibrillation in heart failure. J Am Coll Cardiol. 2013 May 7;61(18):1894-903. doi: 10.1016/j.jacc.2013.01.069. Epub 2013 Mar 7. PMID 23500267